CLINICAL TRIAL: NCT06548724
Title: Patient's Quality of Life and Functional Changes After Fistula Surgery
Status: Recruiting | Type: Observational
Sponsor: Mansoura University Hospital (Other)
Responsible Party: Principal Investigator, Ahmed hossam Elsayed, assistant lecturer of general and Colorectal surgery, Mansoura University Hospital
Other Study IDs: MD.21.08.508
Record Dates: First submitted 2023-11-09; First posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Anal Fistula
Keywords: quality of life; incontinence; preoperative; postoperative
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: assessment of quality of life before and after anal surgery — Preoperatively, the state of continence will be assessed using Wexner Incontinence Score (WIS) . Also, the basal state of quality of life (QoL) will be assessed using a validated disease-specific tool known as Quality of Life in patients with Anal Fistula Questionnaire (QoLAFQ) (Ferrer-Márquez et al., , faecal incontinence quality of life (FIQL)
  Surgical Techniques:
  The selection of surgical technique depends on the type of fistula , patient choice and commitment to guidelines . Follow-up Patients will be followed-up in the outpatient clinic weekly in the first month, then every two weeks in the second month, then at 3, and 6 months postoperatively. The continence state and QoL change will be assessed using QoLAF-Q and GIQLI 3 months and6 months postoperatively.

SUMMARY:
This is a prospective observational study that will monitor the effects of surgery for anal fistula on the patient quality of life using many valid questionnaires

DETAILED DESCRIPTION:
Anal fistulas can be classified as simple or complex. Simple anal fistula includes low trans-sphincteric and intersphincteric fistulas that cross less than 30% of the external sphincter fibers. On the other hand, complex anal fistulas comprise, high trans-sphincteric fistulas, suprasphincteric, extrasphincteric fistulas

Patients with anal fistula often complain of recurrent perianal discharge and pruritus ani. Sometimes recurrent abscesses develop due occlusion of the external opening leading to episodes of fever and exquisite perianal pain. Diagnostic modalities that aid in the diagnosis of anal fistula include fistulography, endorectal ultrasonography, MR Fistulography

While the treatment of simple anal fistula is usually straightforward with fistulotomy being recommended as the first line of treatment ; the management of more complex cases requires more sophisticated treatments aiming to preserve the anal sphincters and to eradicate the fistulous track. Surgery for complex anal fistula includes the placement of Seton, anal advancement flap, laser ablation, fistula plug, and video-assisted anal fistula treatment. There exists a debate about the optimal management of low anal fistula with both fistulectomy and fistulotomy considered as viable options for treatment. Fistulectomy involves complete excision of the fistulous tract, eliminating the risk of missing secondary tracts and providing complete tissue for histopathological examination. On the other hand, fistulotomy involves lay open of the fistulous tract, thus leaving smaller unepithelized wounds, which hastens the wound healing . A recent meta-analysis found no significant difference between both procedures regarding recurrence of anal fistula, yet with accelerated healing time in favor of fistulotomy .Recently, alternative therapies have been employed in the management of cryptogenic anal fistula in an attempt to render the surgery more minimally invasive and to reduce the likelihood of post-operative fecal incontinence .

These treatments have included ligation of the intersphincteric fistula tract (the LIFT procedure) either with or without the deployment of a biosynthetic mesh , or fistula clip closure techniques , and a range of endo-fistula therapies including video-assisted anal fistula treatment (VAAFT) , anal fistula plugs , and a variety of injected biomaterials

, The ''Fistula Laser Closing'' (FiLaCTM) device (Biolitec, Germany) is another endo-fistula management technique . There is few studies assessing the changes in quality of life that occurs after fistula surgery whatever its technique and the aim of this study is t assess the impact of intervention for fistula on patient's quality of life

ELIGIBILITY:
Inclusion Criteria:

* both genders
* Age :between 18-65 years
* cryptoglandular anal fistula
* need intervention

Exclusion Criteria:

- Patients with associated anorectal pathology (anal fissure, hemorrhoids, rectal prolapse, neoplasm, solitary rectal ulcer, inflammatory bowel diseases.)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patient who will be admitted in the General Surgery Department, Colorectal Surgery Unit at Mansura University hospital
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
patient quality of life changes before and after surgery with QoLAF-Q | after 1 and 3 and 6 months
  To Evaluate the impact of the fistula surgery on quality of life , the range range between 14 points which means zero impact on the quality of life and 70 which is the highest impact of anal fistula on the quality of life functional aspect in form of incontinence and quality of life of the patient

SECONDARY OUTCOMES:
the validation of arabic translation of the quesionaire | 3 and 5 months
  The validation of the arabic translation of the questionaire will be done to establish a avalidated form in arabic that can be easily undrestandable for arabic population . it will be done on part of participants in a time frame of 4 to 5 months QoLAF-Q. In addition, postoperative pain, state of continence, manometric changes, operation time, time to healing, and postoperative complications

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura university hospital, Al Mansurah, Dakahlyia, Egypt